CLINICAL TRIAL: NCT04197362
Title: Everyday Activity Shoes: a Quantification of Impact Forces While Walking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to the PI leaving for sabbatical.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, David T. Burke, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB00112113
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Impact Forces
Keywords: activity shoes; forces; torques; cartilage; bones

STUDY DESIGN:
Intervention Model Description: The subjects will be fitted in random order of a pair of ASICS Women's Gel-Venture 6 Running-Shoe, Nike Air Max 270, La Vida+ athletic shoes. Subjects will be pre-assigned randomly to start and continue with specific shoe groups, ultimately exhausting all options.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASICS Women's Gel-Venture 6 Running-Shoe (Experimental): ASICS Women's Gel-Venture 6 Running-Shoe
  Interventions: Other: Evaluation
- Nike Air Max 270 (Experimental): Nike Air Max 270
  Interventions: Other: Evaluation
- La Vida+ (Experimental): La Vida+
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Subjects will be asked to walk across the gait laboratory floor at their self-selected walking speed. They will complete a 3-5 minute warm up period, as it was found to produce stable estimates of kinetic parameter mean values during treadmill activity. The positions of each marker will be recorded through the motion capture system. Ground reaction force will be obtained in real time from the gait laboratory force plates as marker dimensions are recorded. For walking data, two trials of 15 seconds each will be recorded. The second trial will be a redundancy in the setting of potential significant marker dropout.

SUMMARY:
This study aims to directly compare traditional everyday activity shoes (ASICS, Nike) with a shoe created to be flatter, less cushioned, and with less cradling of the foot (OESH shoe).

DETAILED DESCRIPTION:
This study addresses a common question in popular media: what attributes of traditional everyday activity shoes (Nike, New Balance, etc.) make a shoe better or worse. There have been several peer-reviewed studies aimed to answer this by calculating forces and torques at the ankles, knees, and hips while subjects wore shoes with different properties. Such characteristics include heel size, cushioning and side-to-side cradling of the foot. Interestingly, most studies have shown that the lack of a heel, less cushioning, and less cradling of the foot actually improve the biomechanics related to forces and torques, thus decreasing wear and tear on the cartilage and bones of the leg. Wear and tear on cartilage and bone may predispose patients to a bone condition called "osteoarthritis", which is a disease where bones become damaged from rubbing on each other with breakdown of a cartilage "cushion". This study thus aims to directly compare traditional everyday activity shoes (ASICS, Nike) with a shoe created to be flatter, less cushioned, and with less cradling of the foot (OESH shoe).

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-65
* Women who identify as "healthy"
* Women who run or walk for exercise more than three times per week
* Women in the Atlanta, Georgia area

Exclusion Criteria:

* Individuals with history of significant musculoskeletal pathology
* Individuals with musculoskeletal injury at time of testing
* Individuals unable to consent
* Individuals outside of the ages 18-65
* Individuals who are prisoners
* Individuals who do not speak or write in English

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 6 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Differences in torques at the knee comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in forces at the knee comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.

SECONDARY OUTCOMES:
Differences in torques at the bilateral anterior and posterior superior spine comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in forces at the bilateral anterior and posterior superior spine comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in torques at the lateral femoral condyles comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in forces at the lateral femoral condyles comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in torques at the lateral mid-shanks comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in forces at the lateral mid-shanks comparing three study arms | One-time at enrollment, no follow-up day
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in torques at the lateral malleoli comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in forces at the lateral malleoli comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in torques at the second metatarsal heads comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in forces at the second metatarsal heads comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in torques at the heels comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.
Differences in forces at the heels comparing three study arms | One-time at enrollment, no follow-up
  Joint torques and forces will be assessed via 16 markers placed on specified anatomical landmarks of the pelvis and lower extremities as the subjects walk across the gait floor at a self-selected speed. In analysis, joint torques and forces will be calculated through full inverse-dynamic model implementation using the Vicon Plug-In Gait. Differences in torques and peak forces will be calculated by ANOVA along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: David Burke, MD, MA, Principal Investigator — Emory University
Locations (1):
- Emory Rehabilitation Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared